CLINICAL TRIAL: NCT01269658
Title: A Randomized, Multi-Center, Double-Masked, Vehicle-Controlled, Parallel-Group, Safety and Efficacy Study of Azithromycin Ophthalmic Solution, 1% Versus Vehicle for Four Weeks in Subjects With Blepharitis
Brief Title: A Four Week Study of Azithromycin Ophthalmic Solution, 1% Versus Vehicle in Subjects With Blepharitis (P08636)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P08636; P08636
Record Dates: First submitted 2010-12-21; First posted 2011-01-04 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-10

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Azithromycin ophthalmic solution, 1% (Experimental)
  Interventions: Drug: Azithromycin ophthalmic solution, 1%
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Azithromycin ophthalmic solution, 1% — 1 drop twice daily (BID) for the first 2 days and then 1 drop once daily (QD) for the remainder of treatment period (approximately 28 days total)
  Arms: Azithromycin ophthalmic solution, 1%
Drug: Vehicle — 1 drop twice daily (BID) for the first 2 days and then 1 drop once daily (QD) for the remainder of treatment period (approximately 28 days total)
  Arms: Vehicle

SUMMARY:
The purpose of this study is to compare the safety and efficacy of azithromycin ophthalmic solution, 1% versus vehicle over a four-week treatment period in treating the signs and symptoms of subjects with blepharitis and to evaluate the clinical course of the condition under study.

ELIGIBILITY:
Inclusion Criteria:

* Have a current diagnosis of blepharitis
* Have a best corrected visual acuity (BCVA), using corrective lenses if

necessary, in both eyes of at least +0.7

* If female, are non-pregnant or non-lactating

Exclusion Criteria:

* Have a concurrent acute hordeolum (stye) or chalazion
* Have inflammation of the ocular surface
* Have used artificial tears within 48 hours prior to Visit 1 or anticipate

using during the study

* Have had ocular surgery in the past 90 days or will require it during the

study

* Unable to withhold the use of contact lenses during the study
* Have a known hypersensitivity to azithromycin, erythromycin, any other

macrolide antibiotic, or any of the other ingredients in the study

medication

* Have been diagnosed with ongoing glaucoma
* Unable to withhold the use of ocular cosmetic products within 48 hours

prior to Visit 1 and throughout the study

* Have a serious medical condition which could confound study assessments

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Resolution of clinical signs of blepharitis | Day 28

SECONDARY OUTCOMES:
Time to first clinical resolution | Days 7, 14, 21, 28, 42, 56, 70, and 84
Mean and change from baseline for clinical signs of blepharitis | Days 7, 14, 21, 28, 42, 56, 70, and 84
Mean and change from end of dosing for clinical signs of blepharitis | Days 42, 56, 70, and 84
Response to the Blepharitis Symptoms Questionnaire (BSQ) | Days 1, 7, 14, 21, 28, 42, 56, 70, and 84

CONTACTS AND LOCATIONS:
Overall Officials: Charles Johnson, MBChB, Study Chair — Chief Medical Officer